CLINICAL TRIAL: NCT04952402
Title: SARS-CoV-2 Immune Responses After COVID-19 Therapy and Subsequent Vaccine
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: A5404
Record Dates: First submitted 2021-06-28; First posted 2021-07-07 (Actual); Results first posted 2023-05-19 (Actual); Last update posted 2023-05-24 (Actual); Status verified 2023-05

CONDITIONS: Covid19; SARS-CoV2 Infection
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cohort: ACTIV-2/A5401 (Experimental): Participants of the ACTIV-2/A5401 randomized trial who received a select investigational (active) therapy (AZD7442 IM or IV, BRII-196 + BRII 198 IV, SAB 185 (3,840 or 10,240 units/kg) IV, BMS 096414+BMS 986413 subcutaneous, Camostat Oral) or its corresponding comparator (Placebo).
  Interventions: Biological: Study-provided Moderna mRNA-1273 COVID-19 vaccine; Biological: Community-provided Moderna mRNA-1273 COVID-19 Vaccine; Biological: Community-Provided Pfizer-BioNTech BNT162b2 COVID-19 Vaccine
- Cohort: COVID-19 Naïve (Experimental): Participants without known history of prior SARS-CoV-2 infection defined as no known history of any SARS-CoV-2 positive test (non-ACTIV-2/A5401 participants).
  Interventions: Biological: Study-provided Moderna mRNA-1273 COVID-19 vaccine

INTERVENTIONS:
Biological: Study-provided Moderna mRNA-1273 COVID-19 vaccine — Participants received a two-dose series (100 µg (0.5 mL) was administered intramuscularly (IM) at Day 0 and Day 28).
Biological: Community-provided Moderna mRNA-1273 COVID-19 Vaccine — Participants received a two-dose series.
  Arms: Cohort: ACTIV-2/A5401
Biological: Community-Provided Pfizer-BioNTech BNT162b2 COVID-19 Vaccine — Participants received a two-dose series.
  Arms: Cohort: ACTIV-2/A5401

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of mRNA COVID-19 vaccines in:

• People with prior COVID-19 (SARS-CoV-2 infection) who were in the ACTIV-2/A5401 study.

And

• People who have never had COVID-19 (SARS-CoV-2 infection).

DETAILED DESCRIPTION:
A5404 is a phase IV, open-label study. The objective of A5404 is to evaluate how prior investigational therapy for COVID-19 versus comparator (placebo or active comparator) affects vaccine response. The safety of mRNA COVID-19 vaccines is also explored.

Eligible A5404 participants include: Participants of ACTIV-2/A5401 at selected sites who received an investigational therapy or its comparator; and persons without known history of prior SARS-CoV-2 infection defined as no known history of any SARS-CoV-2 positive test (non-A5401 participants). In line with our protocol, for outcome measures related to neutralizing antibodies and adverse events, we further break down the ACTIV-2/A5401 participants into two exposure groups: those who received an active therapy (AZD7442 IM or IV, BRII-196 + BRII 198 IV, SAB 185 (3,840 or 10,240 units/kg) IV, BMS 096414+BMS 986413 subcutaneous) and those who received Camostat Oral or Placebo.

Participants of ACTIV-2/A5401 received study-provided standard dosing of the Moderna mRNA-1273 vaccine, or a community-provided mRNA-based COVID-19 vaccine (e.g., Moderna or Pfizer). Participants in ACTIV-2/A5401 received their mRNA-based COVID-19 vaccine 60-240 days after receiving their last dose of a select ACTIV-2/A5401 investigational therapy, or its comparator. Participants without prior COVID-19 received study-provided standard dosing of the Moderna mRNA-1273 vaccine.

The study closed early to accrual on February 25, 2022 due to slow enrollment. Clarification Memo #1 (dated January 11, 2023) reflects decisions to discontinue follow up at study Day 365 instead of following participants to Day 730 after the first dose of vaccine and to reallocate some secondary outcome measures to exploratory outcome measures.

ELIGIBILITY:
Inclusion Criteria:

* For all participants: Ability and willingness of participant (or legally authorized representative) to provide informed consent prior to initiation of any study procedures.
* For participants who are in, or who have completed, the ACTIV-2/A5401 trial: Receipt of all selected investigational therapy or active comparator/placebo for that therapy at selected sites.
* For participants who are in, or who have completed, the ACTIV-2/A5401 trial and receive study-provided Moderna mRNA-1273 COVID-19 vaccine: Receipt of the last dose of investigational therapy or active comparator/placebo for that therapy ≥30 days and ≤240 days prior to study entry.
* For participants who are in, or who have completed, the ACTIV-2/A5401 trial and have received or will be receiving community-provided mRNA-based COVID-19 vaccine: Receipt of the last dose of investigational therapy or active comparator/placebo for that therapy ≥30 and ≤240 days prior to receipt or planned receipt of the first dose of community-provided vaccine.

Exclusion Criteria:

* For participants who are in, or who have completed, the ACTIV-2/A5401 trial: Self-report of prior receipt of a non-mRNA-based COVID-19 vaccine.
* For participants who are in, or who have completed, the ACTIV-2/A5401 trial: Self-report of receipt of the first dose of an mRNA-based COVID-19 vaccine 140 days or more before A5404 enrollment.
* For participants who are in, or who have completed, the ACTIV-2/A5401 trial: Self-report of a second SARS-CoV-2 infection after the infection that qualified the participant for ACTIV-2/A5401.
* For non-A5401/ACTIV-2 participants: Self-report of receipt of any prior COVID-19 vaccine.
* For non-A5401/ACTIV-2 participants: Known prior history of any SARS-CoV-2-positive test (e.g., PCR test, Nucleic Acid Amplification Test (NAAT), antigen test, serology test).
* For participants who receive study-provided Moderna mRNA-1273 COVID-19 vaccine: Known allergy to any component of the Moderna COVID-19 vaccine.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2021-07-09 (Actual); Primary Completion 2022-02-28 (Actual); Study Completion 2023-01-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Smith, MD, MAS, Study Chair — UCSD Antiviral Research Center
Locations (6):
- United States (6):
  - UCLA CARE Center CRS, Los Angeles, California
  - UCSD Antiviral Research Center CRS, San Diego, California
  - Rush University CRS (Site ID: 2702), Chicago, Illinois
  - Brigham and Women's Hospital Therapeutics Clinical Research Site (BWH TCRS) CRS, Boston, Massachusetts
  - Chapel Hill CRS (Site ID: 3201), Chapel Hill, North Carolina
  - University of Washington AIDS CRS, Seattle, Washington

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie results in the publication, after deidentification.
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 3 months following publication and available throughout period of funding of the AIDS Clinical Trials Group by NIH.
Access Criteria: * With whom? Researchers who provide a methodologically sound proposal for use of the data that is approved by the AIDS Clinical Trials Group.
  * For what types of analyses? To achieve aims in the proposal approved by the AIDS Clinical Trials Group.
  * By what mechanism will data be made available? Researchers may submit a request for access to data using the AIDS Clinical Trials Group "Data Request" form at: https://actgnetwork.org/submit-a-proposal/. Researchers of approved proposals will need to sign an AIDS Clinical Trials Group Data Use Agreement before receiving the data.

REFERENCES:
- See also: The Division of AIDS Table for Grading the Severity of Adult and Pediatric Adverse Events (DAIDS AE Grading Table), corrected Version 2.1, July 2017. — https://rsc.niaid.nih.gov/clinical-research-sites/daids-adverse-event-grading-tables
- See also: Manual for Expedited Reporting of Adverse Events to DAIDS (DAIDS EAE Manual), Version 2.0, January 2010 — https://rsc.niaid.nih.gov/clinical-research-sites/manual-expedited-reporting-adverse-events-daids

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled from July 9, 2021 to December 16, 2021 at six clinical research sites in the U.S.
Pre-assignment Details: For participant flow, ACTIV-2/A5401 participants regardless of the exposure (select active therapy or Camostat or placebo) are considered as one cohort, and COVID-naïve participants are considered as the second cohort.
Period: Overall Study
Arm/Group | Cohort: ACTIV-2/A5401 | Cohort: COVID-19 Naïve
Started | 18 | 25
Completed Two-dose Vaccine Series | 18 | 25
Completed | 17 | 21
Not Completed | 1 | 4
Not completed — Lost to Follow-up | 1 | 3
Not completed — Lack Of Venous Access | 0 | 1

BASELINE CHARACTERISTICS:
Population: All A5404 trial participants. For baseline characteristics, ACTIV-2/A5401 participants regardless of the exposure (select active therapy or Camostat or placebo) are considered as one cohort, and COVID-naïve participants are considered as the second cohort.
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort: ACTIV-2/A5401 | Cohort: COVID-19 Naïve | Total
Number analyzed (Participants) | 18 | 25 | 43
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 35 [28 to 52] | 32 [23 to 42] | 32 [24 to 43]
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 9 | 16 | 25
  Gender Queer | 0 | 1 | 1
  Male | 9 | 8 | 17
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 17 | 26
  Male | 9 | 8 | 17
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 6 | 12
  Not Hispanic or Latino | 12 | 19 | 31
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: Black Or African American | 1 | 18 | 19
  Race: White | 17 | 7 | 24
Body Mass Index [Median (Inter-Quartile Range); unit: kg/m^2] — Population: 8 participants in the ACTV-2/A5401 cohort did not have BMI information collected.
  kg/m^2
    number analyzed (Participants) | 10 | 25 | 35
    (all) | 40 [27 to 46] | 24 [21 to 32] | 27 [21 to 44]

OUTCOME MEASURES:

1. Primary Outcome: Neutralizing Antibody (NAb) Level
Description: NAb level was measured by using both 50% neutralizing dilution titers (ND50) and 80% neutralizing titers (ND80). A higher NAb level corresponds to a stronger immune response. For ND50 values less than lower limit of quantification (LLQ), we impute with 10 (which is ½ LLQ of 20). For ND50 values exceeding the upper limit of quantification (ULQ), we impute with 20,000 (a value suggested by the immunology lab, which is 2 times the ULQ of 10,000). For ND80, we impute similarly with 10 and 20,000. We carry forward the Day 56 NAb measurement if the Day 140 measurement is not reported.
Time Frame: Measured 140 days after the first dose of the vaccine
Population: The analysis population includes all participants who received at least the first dose of an mRNA-based COVID-19 vaccine and who provided a specimen sample at either Day 56 or Day 140 (One COVID-19 naïve participant who was not able to provide specimen at any study visits was excluded).
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Groups:
- ACTIV-2/A5401 Investigational Therapy Except Camostat: Participants of ACTIV-2/A5401 who received an investigational (active) therapy (AZD7442 IM or IV, BRII-196 + BRII 198 IV, SAB 185 (3,840 or 10,240 units/kg) IV or BMS 096414+BMS 986413 subcutaneous).
  Study-provided Moderna mRNA-1273 COVID-19 vaccine: Participants received a two-dose series (100 µg (0.5 mL) was administered intramuscularly (IM) at Day 0 and Day 28).
  Community-provided Moderna mRNA-1273 COVID-19 Vaccine: Participants received a two-dose series.
  Community-Provided Pfizer-BioNTech BNT162b2 COVID-19 Vaccine: Participants received a two-dose series.
- ACTIV-2/A5401 Placebo or Camostat: Participants of ACTIV-2/A5401 who received placebo or Camostat.
  Study-provided Moderna mRNA-1273 COVID-19 vaccine: Participants received a two-dose series (100 µg (0.5 mL) was administered intramuscularly (IM) at Day 0 and Day 28).
  Community-provided Moderna mRNA-1273 COVID-19 Vaccine: Participants received a two-dose series.
  Community-Provided Pfizer-BioNTech BNT162b2 COVID-19 Vaccine: Participants received a two-dose series.
- COVID-19 Naïve: Participants without known history of prior SARS-CoV-2 infection defined as no known history of any SARS-CoV-2 positive test (non-ACTIV-2/A5401 participants)
  Study-provided Moderna mRNA-1273 COVID-19 vaccine: Participants received a two-dose series (100 µg (0.5 mL) was administered intramuscularly (IM) at Day 0 and Day 28).
Arm/Group | ACTIV-2/A5401 Investigational Therapy Except Camostat | ACTIV-2/A5401 Placebo or Camostat | COVID-19 Naïve
Number analyzed (Participants) | 8 | 10 | 24
titer
  50% neutralizing dilution titers (ND50) | 2242.47 [688.55 to 7303.29] | 2695.21 [1005.71 to 7222.88] | 2196.74 [970.88 to 4970.42]
  80% neutralizing dilution titers (ND80) | 888.80 [222.60 to 3548.78] | 972.43 [358.67 to 2636.46] | 794.90 [364.34 to 1734.27]

2. Secondary Outcome: Geometric Mean of Relative Change in Neutralizing Antibody Levels From Pre-vaccine to Post-vaccine
Description: Relative change is defined as the ratio of post-vaccine NAb level/pre-vaccine NAb level. A ratio greater than one indicates an increase of NAb response. For ND50 values less than lower limit of quantification (LLQ), we impute with 10 (which is ½ LLQ of 20). For ND50 values exceeding the upper limit of quantification (ULQ), we impute with 20,000 (a value suggested by the immunology lab, which is 2 times the ULQ of 10,000). For ND80, we impute similarly with 10 and 20,000.
Time Frame: Measured before the first dose of the vaccine, and 56 days after the first dose of the vaccine
Population: The analysis population includes all participants who received at least the first dose of an mRNA-based COVID-19 vaccine and who provided a specimen sample at both Day 0 and Day 56.
Measure: Geometric Mean (95% Confidence Interval); unit: ratio
Arm/Group | ACTIV-2/A5401 Investigational Therapy Except Camostat | ACTIV-2/A5401 Placebo or Camostat | COVID-19 Naïve
Number analyzed (Participants) | 3 | 2 | 21
ratio
  50% neutralizing dilution titers (ND50) | 6.85 [0.05 to 982.60] | 21.63 [0.00 to 1842965.87] | 50.80 [16.66 to 154.86]
  80% neutralizing dilution titers (ND80) | 8.31 [0.01 to 5138.20] | 40.86 [0.18 to 9051.19] | 33.05 [12.19 to 89.59]

3. Secondary Outcome: Proportion of Participants With New Grade 3 or Higher AE, or SAE, or AE Leading to Change or Discontinuation in Vaccine Receipt
Description: An adverse event (AE) is any unfavorable and unintended sign, symptom, or diagnosis that occurs in a study participant during the conduct of the study REGARDLESS of the attribution. A serious adverse event (SAE) is defined as any untoward medical occurrence that results in death; is life-threatening; requires inpatient hospitalization or prolongation of existing hospitalization; results in persistent or significant disability/incapacity; is a congenital anomaly/birth defect; is an important medical event that may not be immediately life-threatening or result in death or hospitalization but may jeopardize the patient or may require intervention to prevent one of the other outcomes listed in the definition above.
  Adverse events are graded on a scale from 1-5: 1=mild, 2=moderate, 3=severe, 4=life-threatening, 5=death. AE grading was per Division of AIDS Table for Grading the Severity of Adult and Pediatric Adverse Events (DAIDS AE Grading Table V2.1).
Time Frame: From first dose of the vaccine through 140 days after the first dose of the vaccine
Population: The analysis population includes all participants who received at least the first dose of an mRNA-based COVID-19 vaccine.
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | ACTIV-2/A5401 Investigational Therapy Except Camostat | ACTIV-2/A5401 Placebo or Camostat | COVID-19 Naïve
Number analyzed (Participants) | 8 | 10 | 25
proportion of participants | 0.13 [0.00 to 0.53] | 0.00 [0.00 to 0.31] | 0.00 [0.00 to 0.14]

4. Secondary Outcome: Number of Participants With Grade 1 or Higher Allergic Reaction
Description: Adverse events are graded on a scale from 1-5: 1=mild, 2=moderate, 3=severe, 4=life-threatening, 5=death. AE grading was per Division of AIDS Table for Grading the Severity of Adult and Pediatric Adverse Events (DAIDS AE Grading Table V2.1).
Time Frame: From first dose of the vaccine through 56 days after the first dose of the vaccine
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | ACTIV-2/A5401 Investigational Therapy Except Camostat | ACTIV-2/A5401 Placebo or Camostat | COVID-19 Naïve
Number analyzed (Participants) | 8 | 10 | 25
Participants | 0 | 0 | 0

5. Secondary Outcome: Proportion of Participants With Grade 2 or Higher Injection Site Reaction
Description: as for outcome 4
Time Frame: From first dose of the vaccine through 56 days after the first dose of the vaccine
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | ACTIV-2/A5401 Investigational Therapy Except Camostat | ACTIV-2/A5401 Placebo or Camostat | COVID-19 Naïve
Number analyzed (Participants) | 8 | 10 | 25
proportion of participants | 0.00 [0.00 to 0.37] | 0.10 [0.00 to 0.45] | 0.00 [0.00 to 0.16]

6. Secondary Outcome: Geometric Mean of Relative Change in Neutralizing Antibody Levels From Pre-vaccine to Post-vaccine by Received Vaccine
Description: Relative change is defined as the ratio of post-vaccine NAb level/pre-vaccine NAb level by received vaccine, i.e., Moderna mRNA-1273 versus Pfizer-BioNTech BNT162b2. A ratio greater than one indicates an increase of NAb response for those on Moderna mRNA-1273 versus Pfizer-BioNTech BNT162b2. For ND50 values less than lower limit of quantification (LLQ), we impute with 10 (which is ½ LLQ of 20). For ND50 values exceeding the upper limit of quantification (ULQ), we impute with 20,000 (a value suggested by the immunology lab, which is 2 times the ULQ of 10,000). For ND80, we impute similarly with 10 and 20,000.
Time Frame: Measured before the first dose of the vaccine, and 56 days after the first dose of the vaccine
Population: The analysis population includes all participants who received at least the first dose of an mRNA-based COVID-19 vaccine and who provided a specimen sample at both Day 0 and Day 56. None of the participants who received Pfizer-BioNTech BNT162b2 COVID-19 vaccine provided a specimen sample at both Day 0 and Day 56.
Measure: Geometric Mean (95% Confidence Interval); unit: ratio
Groups:
- Participants Who Received Study or Community-provided Moderna mRNA-1273 COVID-19 Vaccine: Participants from the ACTIV-2/A5404 cohort or the COVID-19 Naïve cohort.
  Study-provided Moderna mRNA-1273 COVID-19 vaccine: Participants received a two-dose series (100 µg (0.5 mL) was administered intramuscularly (IM) at Day 0 and Day 28).
  Community-provided Moderna mRNA-1273 COVID-19 Vaccine: Participants received a two-dose series.
- Participants Who Received Community-provided Pfizer-BioNTech BNT162b2 COVID-19 Vaccine: Participants from the ACTIV-2/A5404 cohort.
  Community-Provided Pfizer-BioNTech BNT162b2 COVID-19 Vaccine: Participants received a two-dose series.
Arm/Group | Participants Who Received Study or Community-provided Moderna mRNA-1273 COVID-19 Vaccine | Participants Who Received Community-provided Pfizer-BioNTech BNT162b2 COVID-19 Vaccine
Number analyzed (Participants) | 26 | 0
ratio
  50% neutralizing dilution titers (ND50) | 37.75 [14.48 to 98.43] |
  80% neutralizing dilution titers (ND80) | 28.65 [12.05 to 68.13] |

7. Other Pre Specified Outcome: CD4+ T Cell Response to SARS-CoV-2 Spike Protein
Description: Team re-prioritized the analysis of secondary objectives due to limited accrual and moved this outcome to exploratory.
Time Frame: At the visit 56 days after the first dose of the vaccine
Reporting Status: Not Posted

8. Other Pre Specified Outcome: CD8+ T Cell Response to SARS-CoV-2 Spike Protein
Description: Team re-prioritized the analysis of secondary objectives due to limited accrual and moved this outcome to exploratory.
Time Frame: At the visit 56 days after the first dose of the vaccine
Reporting Status: Not Posted

9. Other Pre Specified Outcome: IgG Serologic Response to SARS-CoV-2 Spike Protein at Receptor Binding Domain (RBD) and N Terminal Domain (NTD) and Matrix (M) Protein.
Description: Team re-prioritized the analysis of secondary objectives due to limited accrual and moved this outcome to exploratory.
Time Frame: At the visit 56 days after the first dose of the vaccine
Reporting Status: Not Posted

10. Other Pre Specified Outcome: Flow Cytometry of PBMC for Markers of Exhaustion on B and T Cells
Description: Team re-prioritized the analysis of secondary objectives due to limited accrual and moved this outcome to exploratory.
Time Frame: At study entry/Day 0 and 56 days after the first vaccine dose.
Reporting Status: Not Posted

11. Other Pre Specified Outcome: IgM Serologic Response to SARS-CoV-2 Spike Protein at Receptor Binding Domain (RBD) and N Terminal Domain (NTD) and Matrix (M) Protein.
Description: Team re-prioritized the analysis of secondary objectives due to limited accrual and moved this outcome to exploratory.
Time Frame: At the visit 56 days after the first dose of the vaccine
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: From study entry through 1 year after receiving the first dose of vaccine.
Description: Any unfavorable/unintended sign/lab finding/symptom/dx during the study REGARDLESS of attribution inc. any occurrence new in onset/aggravated in severity/frequency from baseline. SAE/EAEs should also be entered into the DAIDS Adverse Experience Reporting System. AE grading was per Division of AIDS Table for Grading the Severity of Adult and Pediatric Adverse Events (V2.1).
Arm/Group | ACTIV-2/A5401 Investigational Therapy Except Camostat | ACTIV-2/A5401 Placebo or Camostat | COVID-19 Naïve
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/10 | 0/25
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/10 | 0/25
Other Adverse Events (participants affected / at risk) | 2/8 | 8/10 | 7/25
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | ACTIV-2/A5401 Investigational Therapy Except Camostat (N=8) | ACTIV-2/A5401 Placebo or Camostat (N=10) | COVID-19 Naïve (N=25)
Peptic ulcer (Gastrointestinal disorders) | 0 | 1 | 0
Fatigue (General disorders) | 0 | 1 | 0
Inflammation (General disorders) | 0 | 1 | 0
Injection site pain (General disorders) | 0 | 1 | 0
Peripheral swelling (General disorders) | 0 | 1 | 0
Acute sinusitis (Infections and infestations) | 0 | 1 | 0
COVID-19 (Infections and infestations) | 1 | 2 | 2
Epididymitis (Infections and infestations) | 0 | 1 | 0
Pharyngitis streptococcal (Infections and infestations) | 0 | 1 | 0
Suspected COVID-19 (Infections and infestations) | 0 | 1 | 0
Hand fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Joint stiffness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Headache (Nervous system disorders) | 0 | 1 | 2
Lumbar radiculopathy (Nervous system disorders) | 0 | 0 | 1
Tremor (Nervous system disorders) | 0 | 1 | 0
Anxiety disorder (Psychiatric disorders) | 1 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 1 | 0
Breast mass (Reproductive system and breast disorders) | 0 | 1 | 0
Vulvovaginal dryness (Reproductive system and breast disorders) | 0 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Rhinitis perennial (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Alopecia areata (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Hypertension (Vascular disorders) | 0 | 0 | 1

LIMITATIONS AND CAVEATS:
The study closed early to accrual due to difficulty enrolling participants. Therefore the sample size is very small and precision is limited.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (5):
  • Study Protocol: Protocol Version 3.0 (2022-11-30): https://cdn.clinicaltrials.gov/large-docs/02/NCT04952402/Prot_000.pdf
  • Study Protocol: Clarification Memo (2023-01-11): https://cdn.clinicaltrials.gov/large-docs/02/NCT04952402/Prot_001.pdf
  • Study Protocol: Letter of Amendment #1 (2021-07-12): https://cdn.clinicaltrials.gov/large-docs/02/NCT04952402/Prot_002.pdf
  • Statistical Analysis Plan (2023-01-27): https://cdn.clinicaltrials.gov/large-docs/02/NCT04952402/SAP_003.pdf
  • Informed Consent Form (2022-11-30): https://cdn.clinicaltrials.gov/large-docs/02/NCT04952402/ICF_004.pdf